CLINICAL TRIAL: NCT01832376
Title: Treatment of Calcific Tendinitis by Ultrasound-guided Needle Lavage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vestre Viken Hospital Trust (Other)
Responsible Party: Principal Investigator, Stefan Moosmayer, MD, PhD, Vestre Viken Hospital Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012/773
Record Dates: First submitted 2013-04-08; First posted 2013-04-16 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Calcific Tendinitis
Keywords: Calcific tendinitis; Shoulder; Needle lavage; Ultrasound-guided

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ultrasound guided needle lavage (Experimental): Ultrasound guided needle lavage
  Interventions: Procedure: Ultrasound guided needle lavage

INTERVENTIONS:
Procedure: Ultrasound guided needle lavage — A 18-gauge needle connected to a 5 ml syringe with 4 ml of saline solution will be used to puncture the calcification with freehand technique and under constant sonographic monitoring. With the tip of the needle placed in the center of the deposit, the calcification will be flushed. If backflow of calcific material can be identified in the syringe, lavage of the deposit will be performed by successive propulsion and aspiration with the syringe plunger. In cases where no material can be extracted, repeated perforation of the deposit will be performed to possibly initiate or accelerate spontaneous resorption.
  Other Names: Barbotage

SUMMARY:
Study population: Subjects with long standing symptoms from calcific tendonitis, non-responsive to other forms of conservative treatment

Study method: A cohort of 50 patients with symptomatic calcific tendonitis will be treated by ultrasound-guided needle lavage. At baseline all study subjects will be assessed by clinical examination, imaging of the shoulder by x-ray and sonography and by the self-report section of the American Shoulder and Elbow Surgeons score (ASES). Follow-up will be performed after 1 and 4 weeks (score only), 3 (clinical, score, ultrasound, x-ray), 6 and 12 months (score only), and after 24 months (clinical, score, ultrasound, x-ray). Patients with insufficient treatment effect will be offered physiotherapy, re-lavage or surgical treatment by acromioplasty.

Purpose of the study: The investigators want to find out

* if shoulder function, measured by a shoulder score, will increase during follow-up
* how much of the calcific material can be aspirated (in ml)
* to which extend the calcific deposit disappears on x-rays and sonographic images
* how many patients will need surgical treatment

ELIGIBILITY:
Inclusion Criteria:

* Shoulder pain for at least 6 months, localised laterally on the upper humerus
* Painful arc
* Positive Hawkins test and/or Neers tegn for impingement
* Calcific deposit of >= 5 mm on shoulder x-ray, verified on sonography with a localisation in the supraspinatus or infraspinatus tendon

Exclusion Criteria:

* The presence of other local or systemic diseases affecting shoulder function like arthritis, inflammatory arthropathy or instability
* Symptoms from a cervical root syndrome
* Sonographic or MRI findings for a rotator cuff tear
* Earlier surgery in the study shoulder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-06; Primary Completion 2016-02 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
The self-report section of the American Shoulder and Elbow Surgeons score (ASES) | Baseline and 24 months
  The self-report section of the American Shoulder and Elbow Surgeons score (ASES) consists of two equally weighted parts for pain and shoulder function, each contributing 50 points to a maximum score of 100. Pain measurement is performed on a 10 cm visual analogue scale divided into 1 cm increments. Shoulder function is measured by classifying 10 activities of daily living on a four-point ordinal scale. Change in points on the ASES scale from baseline to 24 month follow-up is the primary outcome measure of our study.

SECONDARY OUTCOMES:
Number of patients who need operative treatment during follow-up | Baseline to 24 months

OTHER OUTCOMES:
Size of the calcific deposit as determined on X-rays of the affected shoulder | Baseline to 3 months and 24 months
  Standardized X-rays of the shoulder are taken at baseline, 3 and 24 month follow-up and the size of the calcific deposits will be measured and compared between examinations

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Moosmayer, MD, PhD, Principal Investigator — Martina Hansens Hospital, Sandvika, Norway
Locations (1):
- Martina Hansens Hospital, Sandvika, Norway

REFERENCES:
- [Result] Moosmayer S and Aasen IB. Ultrasound- Guided Percutaneous Needle Treatment and Steroid Injection for Calcific Tendinopathy of the Shoulder: Can the Orthopedic Surgeon do it?. M J Orth. 3(1): 020, 2018.
- See also: Study publication, open access — http://www.mathewsopenaccess.com/PDF/orthopedics/M_J_Orth_3_1_020.pdf